CLINICAL TRIAL: NCT00882466
Title: Phase 4 Study of the Effect of Human Recombinant Erythropoietin at the Time of Reperfusion in Patients With Acute Myocardial Infarction
Brief Title: The Effect of Erythropoietin at the Time of Reperfusion in Acute Myocardial Infarction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Dong-Ju Choi, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPO in AMI
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2009-04

CONDITIONS: Acute Myocardial Infarction
Keywords: erythropoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI only (No Intervention): primary PCI only
- EPO (Experimental)
  Interventions: Drug: human recombinant erythropoietin

INTERVENTIONS:
Drug: human recombinant erythropoietin — intravenous bolus injection of EPO (50unit/kg)
  Arms: EPO

SUMMARY:
The purpose of this study is to investigate the effect of intravenous human recombinant erythropoietin on the reperfusion injury at primary percutaneous coronary intervention in patients with acute myocardial infarction.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction <12hr
* Age >18yrs
* First myocardial infarction
* culprit lesion : proximal to mid left anterior descending artery
* Baseline coronary flow : TIMI Grade 0~1

Exclusion Criteria:

* Patients with previous myocardial infarction
* History of thrombotic complication
* History of cerebral infarction
* Uncontrolled hypertension
* Increased hemoglobin level >17g/dL
* Patients with mechanical valve
* Cardiogenic shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2008-05; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Creatinine kinase (CK), creatinine kinase-MB (CK-MB) | 4hr, 8hr, 12hr, 24hr, 48hr, 72hr

SECONDARY OUTCOMES:
Infarct size assessed by cardiac MRI | day 4

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju Choi, MD,PhD, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, South Korea

REFERENCES:
- [Derived] Suh JW, Chung WY, Kim YS, Kim KI, Jeon EJ, Cho YS, Youn TJ, Chae IH, Kim CH, Choi DJ. The effect of intravenous administration of erythropoietin on the infarct size in primary percutaneous coronary intervention. Int J Cardiol. 2011 Jun 2;149(2):216-220. doi: 10.1016/j.ijcard.2010.02.002. Epub 2010 Mar 2. PMID 20199815